CLINICAL TRIAL: NCT07356362
Title: The Effectiveness of High-power Laser Therapy in the Treatment of Notalgia Paresthetica: A Randomised Controlled Study.
Brief Title: High-power Laser Therapy for Notalgia Paresthetica.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uşak University (Other)
Collaborators: Balikesir University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AYK&ES&NS notalgia
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Notalgia Paresthetica
Keywords: Laser Therapy; Pain; Itching; Discopathy; Neuropathy
MeSH Terms: conditions — Pain; Pruritus

STUDY DESIGN:
Intervention Model Description: This is a parallel assignment. It is a controlled trial. Design: This is a prospective randomised study. It is assessor-blinded. It is two-arm parallel-group.
Who Masked: Outcomes Assessor
Masking Description: Assessors will be blinded. The clinician conducting the outcome assessments will be unaware of group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group: High-Power Laser Therapy group (Experimental): Methodology for application, method for scanning, the laser probe will be shifted gradually and without interruption over the whole length of the LFCN (from just the medial and inferior aspects of the ASIS, distally along the thigh).
  Interventions: Device: High-power laser
- Sham Laser Group (Sham Comparator): The procedure is the same as Group 1, but without the therapeutic energy emitted by the sham laser applicator. The device will make a beeping sound and show a display as if it is functioning.
  Interventions: Other: Sham Laser

INTERVENTIONS:
Device: High-power laser — Wavelength: 1064 nm Output power: 10 W (continuous wave) Spot size: 8 cm² Energy density: 100 J/cm² per session Application technique: The laser probe will be applied using a scanning technique over the affected dermatomal area and the corresponding paravertebral muscles from T2 to T6 levels.
  Treatment duration: 10 minutes per session Frequency: 3 sessions per week for 4 weeks (total 12 sessions)
  Arms: Experimental Group: High-Power Laser Therapy group
Other: Sham Laser — Participants will receive identical positioning and procedures as the experimental group, using the same laser device with a sham applicator that emits no therapeutic energy. The device will display active operation and produce typical sounds to maintain blinding.
  Arms: Sham Laser Group

SUMMARY:
A non-invasive modality for the management of neuromusculoskeletal pain conditions that has emerged as a compelling option is high-power laser therapy (HPLT). The pathophysiology of notalgia paresthetica (NP) is treated uniquely by HPLT, which targets both the presumed muscular component of nerve entrapment and the resultant neuropathic symptoms. The main goal of this study, which is randomised, controlled and blinded by assessors, is to find out how well High-Power Laser Therapy (HPLT) works as an extra treatment to standard care in reducing itching, pain and improving quality of life for patients with long-term nerve pain.

DETAILED DESCRIPTION:
Notalgia Paresthetica (NP) is a sensory mononeuropathy characterized by a well-circumscribed area of pruritus, paresthesia, burning pain, and hyperpigmentation on the medial aspect of the scapular and infrascapular regions. The condition results from the entrapment or compression of the posterior rami of the thoracic spinal nerves T2 through T6 as they traverse through the multifidus spinae muscle, making a sharp turn to penetrate the fascia of the back muscles. This anatomical vulnerability creates a predisposition to nerve irritation, leading to the characteristic symptoms. NP is often chronic and recalcitrant to treatment, with significant negative impacts on sleep, daily activities, and quality of life.

The current management of NP is challenging and often unsatisfactory. First-line treatments typically include topical agents such as capsaicin cream, topical anesthetics, or corticosteroids to alleviate localized symptoms. For more persistent cases, systemic medications like gabapentinoids or tricyclic antidepressants may be employed, though their efficacy is variable and side effects can be limiting. Interventional procedures, including trigger point injections with anesthetics and corticosteroids, or botulinum toxin A injections, have shown promise by targeting the underlying muscular entrapment. However, the evidence base for these interventions remains limited, consisting largely of case reports and small series, highlighting a significant gap in the availability of effective, non-invasive, and well-tolerated therapeutic options.

High-Power Laser Therapy (HPLT) has emerged as a compelling non-invasive modality for the management of neuromusculoskeletal pain conditions. Operating at power outputs typically between 1 and 15 Watts, HPLT utilizes wavelengths (e.g., 980 nm, 1064 nm) that provide deep tissue penetration, reaching the affected neurovascular structures beneath the thick paraspinal musculature. The therapeutic mechanisms of HPLT are multifactorial, combining significant photothermal effects with photobiomodulation. These include deep tissue analgesia, reduction of inflammation and edema, relaxation of hypertonic muscles, enhanced microcirculation, and stimulation of nerve repair processes. By targeting both the presumed muscular component of nerve entrapment and the resultant neuropathic symptoms, HPLT presents a uniquely suited, non-pharmacological intervention for the pathophysiology of NP.

Despite the growing body of evidence supporting HPLT for various entrapment neuropathies, such as meralgia paresthetica, its application specifically for Notalgia Paresthetica remains largely unexplored. A rigorous, controlled investigation is necessary to determine its clinical value and establish it as a viable treatment option.

Aim of the Study

The primary aim of this randomized, sham-controlled, assessor-blinded study is to investigate the efficacy of High-Power Laser Therapy (HPLT) as an adjunct to standard care on pruritus intensity, pain, and quality of life in patients with chronic Notalgia Paresthetica.

This study hypothesize that patients receiving active HPLT will demonstrate significantly greater reduction in pruritus and pain scores, alongside greater improvement in quality of life, compared to those receiving a sham laser procedure.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-75 years
* Clinical diagnosis of unilateral Notalgia Paresthetica for at least 3 months
* Presence of characteristic symptoms (pruritus, paresthesia, and/or burning pain) in the typical T2-T6 dermatomal distribution
* A minimum score of 4 on the Numeric Rating Scale (NRS) for pruritus intensity
* Presence of hyperpigmentation in the affected area

Exclusion Criteria:

* - Secondary causes of symptoms (e.g., spinal pathology, herpes zoster, renal failure)
* Previous spinal surgery in the thoracic region
* Coagulopathy or use of anticoagulant medication
* Skin diseases or infections in the treatment area
* Pregnancy or lactation
* Cognitive impairment affecting ability to complete questionnaires
* Previous treatment with botulinum toxin in the affected area within 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-27 (Estimated); Primary Completion 2026-10-23 (Estimated); Study Completion 2026-11-12 (Estimated)

PRIMARY OUTCOMES:
Pain screening with PainDETECT | Baseline, 3rd week, 3rd months
  PainDETECT screening questionnaire: PainDETECT is a simple, easy to use screening questionnaire. The questionnaire consists of 9 items and is completed by the patient (no clinical examination is required). There are 7 weighted sensory descriptor items (never to very strongly) and 2 items relating to spatial and temporal pain characteristics. A total score of 19 or more is indicative of likely neuropathic pain.

SECONDARY OUTCOMES:
Pruritus Intensity | Baseline, 3rd week, 3rd months
  Measured using the Numeric Rating Scale (NRS) for pruritus. It can be interpreted as follows:
  Score 0 = no pruritus Score < 3 = mild pruritus Score ≥3<7 = moderate pruritus Score ≥7<9 = severe pruritus Score ≥9 = very severe pruritus

CONTACTS AND LOCATIONS:
Overall Officials: Ender Y Salbas, Asst. Prof., Study Chair — University of Balikesir